CLINICAL TRIAL: NCT04204395
Title: Efficacy of Peanut Ball Usage on Labor Pain, Support and Control, Anxiety, and Labor Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201910010
Record Dates: First submitted 2019-12-02; First posted 2019-12-19 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2019-11

CONDITIONS: Labor Pain
Keywords: Peanut Ball; Labor Pain; Support and Control; Anxiety; Labor Duration
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): When complete the admission process, the caregiver will give a peanut ball to perform, besides the routine health brochure.
  The participants will be at independent compartment.
  Interventions: Device: Peanut Ball
- Control group (No Intervention): Take the routine health brochure. The participants will be at independent compartment.

INTERVENTIONS:
Device: Peanut Ball — The participants in the experimental group will use the peanut ball at least every 2 hours, 30-minute usage for each time. More frequency will be available. Then, the participants will stop using the peanut ball when cervical os is dilated and effaced, may be ready to push.
  Arms: Experimental group

SUMMARY:
*Primary: To compare the control group, women in the experimental group will have lower level of labor pain after the intervention of peanut ball usage.

*Secondary: To compare the control group, women in the experimental group will have higher level of support and control after the intervention of peanut ball usage; To compare the control group, women in the experimental group will have lower level of anxiety after intervention of peanut ball usage; To compare the control group, women in the experimental group will have shorter duration of labor after intervention of peanut ball usage.

DETAILED DESCRIPTION:
We will ask the participants to join this research on the department of obstetric outpatient department, and give the consent form to sign. Then we will allocate the participant into the experiment group or the control group, furthermore, we will give the sheet which includes the information about peanut ball usage, like the destination, method, position, duration, and quick response code of the video.

When they finish the admission process in the delivery room, we will give the peanut ball to the participants who is in the experimental group, and the participants of the control group will receive the routine care of delivery room.

ELIGIBILITY:
Inclusion Criteria:

1. vaginal birth;
2. pregnant women at ≥3 6 weeks of gestation;
3. greater than 20 years old of age;
4. no major obstetric or medical complications;
5. singleton pregnancy;
6. the partner will be accompanied during the labor;
7. cervical dilation is less than 5 cm;
8. able to listen, speak, read and write in Chinese;
9. complete the informed consent form.

Exclusion Criteria:

1. emergency cesarean section;
2. diagnosed with metal disease or drug abuser;
3. complicated with abnormality during labor.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changed perception of Pain | The baseline will be assessed when the cervical dilation is during 0 to 3 centimeters. The three post-tests will be assessed when 30 minutes after each intervention, and cervical dilation is during 5 to 7 centimeters, and during 8 to 10 centimeters.
  Perception of Pain assessed by Visual analogue scale for pain(VAS-P). Range of the VAS-P score is 0 to 10, higher scores means worse outcome.

SECONDARY OUTCOMES:
Changed perception of Support and Control in Birth | The baseline will be assessed when the cervical dilation is during 0 to 3 centimeters. The post-test will be assessed within 24 hours after delivery.
  Perception of Support and Control assessed by Chinese version support and control scale in birth(C-SCIB). The range of the score is from 33 to 165, higher score means better outcome.
Changed perception of anxiety | The baseline will be assessed when the cervical dilation is during 0 to 3 centimeters. The three post-tests will be assessed when 30 minutes after each intervention, and cervical dilation is during 5 to 7 centimeters, and during 8 to 10 centimeters.
  Perception of anxiety assessed by Visual analogue scale for anxiety(VAS-A). Range of the score is 0 to 10, higher scores means worse outcome.
Duration of labor | within 24 hours after delivery
  Duration of labor from Medical record sheet
Changed trajectory of Heart Rate Variability | The baseline will be assessed when the cervical dilation is during 0 to 3 centimeters. The three post-tests will be assessed when 30 minutes after each intervention, and cervical dilation is during 5 to 7 centimeters, and during 8 to 10 centimeters.
  Heart Rate Variability assessed by Heart Rate Variability Device which indicates the sympathetic nervous system status.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, PhD., Study Director — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No